CLINICAL TRIAL: NCT01296308
Title: Effectiveness of a Complementary and Integrative Therapy in Diabetic Neuropathy Patients.
Brief Title: Complementary and Integrative Therapy for Diabetic Neuropathy
Acronym: CIT-DN
Status: Completed | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, MSc, Universität Duisburg-Essen
Other Study IDs: 10-4517
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Neuropathy
Keywords: Diabetes Mellitus, Type 2; Diabetic Neuropathy; Complementary Medicine; Alternative Medicine; Integrative Medicine; Quality of Life; Quantitative Sensory Testing
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- type 2 diabetics with neuropathy
  Interventions: Other: inpatient integrative treatment

INTERVENTIONS:
Other: inpatient integrative treatment — two weeks inpatient integrative therapy: conventional medicine, traditional European and Chinese medicine (TCM), mind-body medicine, physical therapy, lifestyle modification program: nutrition advices, stress management, exercise training

SUMMARY:
Despite the long tradition of complementary and alternative medicine (CAM) therapies there are hardly any interventional trials on type 2 diabetes mellitus. Hence this pilot study aims to investigate the influence of a two weeks integrative inpatient therapy on the quality of life in 50 patients suffering from diabetic neuropathy. Integrative treatment includes aspects of conventional and traditional European and Chinese medicine, mind-body medicine, physical therapy and lifestyle modification (nutrition advices, stress management and exercise training). The observational design intends four measurement points: tree months before (T0), directly before (T1), directly after treatment (T2) and three months follow-up (T3). The subjective evaluation of the neuropathy-related quality of life was combined with neurophysiologic instruments (QST), to measure neuropathic symptoms. Also pain intensity, locus of control, interpretation of illness, coping style, anxiety/depression, life satisfaction and several biomarkers (HbA1c, ABI, WHR and BMI) are measured. In addition a qualitative interview should give a view to patient perspective of therapy process.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* diabetes mellitus type 2

Exclusion Criteria:

* diabetes mellitus type 1
* pregnancy
* oncologic diseases
* systemic neurological diseases
* other induced neuropathy (radicular, s/p alcohol abuse, chemotherapy-induced)
* other severe psychiatric or somatic comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Neuropathy-related Quality of Life (QOL-DN) | at T2
  Norfolk Quality of Life Questionnaire (Vinik et al. 2008)
Neuropathy-related Quality of Life (QOL-DN) | at T3
  Norfolk Quality of Life Questionnaire (Vinik et al. 2008)

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST) | at T2 and T3
  * Thermal detection thresholds (CDT, WDT), thermal pain thresholds (CPT, HPT) and paradoxical heat sensations (PHS)
  * Mechanical detection threshold (MDT), mechanical pain threshold (MPT), mechanical pain sensitivity (MPS), dynamic mechanical allodynia (ALL) and wind-up ratio (WUR)
  * Vibration detection threshold (VDT)
  * Pressure pain threshold (PPT) (Rolke et al. 2006)
Pain intensity (VAS) | at T2 and T3
  100mm Visual Analogue Scale
Control Beliefs (MHLC / short form) | at T2 and T3
  Short form of the Multidimensional Helath Locus of Control Scale (Hasenbring 1988)
Interpretation of Illness (IIQ) | at T2 and T3
  Interpretation of Illness Questionnaire (Büssing et al. 2009)
Coping Style (AKU) | at T2 and T3
  Short form of the Adaptive Coping with Disease Questionnaire (Büssing et al. 2010)
Anxiety and Depression (HADS) | at T2 and T3
  Hospital Anxiety and Depression Scale (Herrmann et al. 1995)
Life Satisfaction (SWLS) | at T2 and T3
  Satisfaction with Life Scale (Diener et al. 1995)
Blood sugar Level (HbA1c) | at T2 and T3
Waist-to-Hip Ratio (WHR) and Body Mass Index (BMI) | at T2 and T3

CONTACTS AND LOCATIONS:
Overall Officials: Gustav J. Dobos, Prof. MD, Principal Investigator — University of Duisburg-Essen
Locations (1):
- Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany